CLINICAL TRIAL: NCT04749836
Title: Registry of His Bundle, Bachmann Bundle and Left Bundle Branch Area Pacing for Various Pacing Indications
Brief Title: Outcomes and Safety of Various Conduction System Pacing Methods
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, David Žižek, MD, PhD, Head of electro-stimulation program, University Medical Centre Ljubljana
Other Study IDs: Conduction pacing Registry
Record Dates: First submitted 2021-02-04; First posted 2021-02-11 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: AV Block; Bundle-Branch Block; Atrial Fibrillation Rapid
Keywords: His bundle pacing; Left bundle branch area pacing; Bachmann bundle pacing
MeSH Terms: conditions — Atrioventricular Block; Bundle-Branch Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: His bundle pacing implantation, Left bundle branch area pacing implantation, Bachmann bundle pacing — Different active fixation leads and the dedicated delivery sheaths are introduced via standard transvenous approach under fluoroscopic guidance. His bundle potential mapping is performed in a unipolar setting with the use of the electrophysiological system for His bundle pacing. After localizing the His bundle potential, the pacing is attempted before the lead fixation to confirm HB capture. The lead is then screwed into position. Acute HBP threshold ≤ 2.5V at 1ms is considered acceptable. On the other hand, the initial site for LBBP is approximately 1-1.5 cm distal to the HBP lead position in the RV septum along the line between the HBP site and RV apex in the right anterior oblique (30°) fluoroscopic view. Bachmann bundle pacing (upper atrial septum) will be performed with the J-stylet modification technique or with specialized catheter method using the SelectSecure active fixation lead.
  Stepwise approach for conduction pacing will also be tested.

SUMMARY:
The aim of this study is to evaluate safety and clinical outcomes after different pacing approaches of conduction system pacing in a prospective registry.

DETAILED DESCRIPTION:
In comparison with right ventricular pacing-induced electromechanical dyssynchrony, conduction system pacing is providing physiological pacing via His-Purkinje activation. Current approaches include His bundle (HBP), left bundle branch area pacing (LBBAP), and Bachmann bundle pacing. In addition, HBP and LBBAP enable correction of underlying proximal bundle branch block, consequently improving the ventricular activation time and narrowing the QRS. Furthermore, atrial activation can be improved with direct Bachmann bundle stimulation. However, the data regarding long-term performance and safety of these physiological approaches in various clinical scenarios is scarce.

With this registry, the investigators would like to obtain real-world data regarding the feasibility and safety of this physiological pacing approaches in various pacing indications and their implementation in routine clinical practice.

Implant success rate, specific implant characteristics, procedural complications, electrical parameters and clinical outcomes will be analyzed at implantation, 1-3 months after inclusion and every 6 months thereafter. Minimal follow-up will be 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Class I and II indications for permanent pacing
* Atrial fibrillation with uncontrolled ventricular rate for pace and ablate strategy
* Bundle branch block correction for HF patients
* Patients with prolonged PR interval and dromotropathy

Ages: 5 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All comers with pacing indication as described in eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-04 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Acute and long-term implant success rate | through study completion, an average of 2 years
  Ventricular activation occurring over the conduction system with acceptable pacing threshold

SECONDARY OUTCOMES:
Pacing parameters | peri-procedural
  Capture threshold, R waves, lead impedance, QRS morphology
Stepwise approach of pacing modes | peri-procedural
  Proportion of patients with HBP as a first option and LBBA as a fist option
Pacing lead stability | through study completion, an average of 2 years
  Lead threshold fluctuation
Heart failure hospitalisation | through study completion, an average of 2 years
  Incidence of heart failure hospitalizations after device implantation
Echocardiographic measurements | through study completion, an average of 1 year
  Assessment of cardiac function
Procedural characteristics | peri-procedural
  Total procedure and fluoroscopy time in minutes

CONTACTS AND LOCATIONS:
Overall Officials: David Žižek, Assist. Prof., Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- University Medical Centre Ljubljana - Cardiology department, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Das A, Banerjee S, Mandal SC. A simple method for Bachmann's bundle pacing with indigenous modification of J-stylet. Indian Heart J. 2016 Sep-Oct;68(5):678-684. doi: 10.1016/j.ihj.2015.10.299. Epub 2016 Jan 11. PMID 27773407
- [Background] Sharma AD, Rizo-Patron C, Hallstrom AP, O'Neill GP, Rothbart S, Martins JB, Roelke M, Steinberg JS, Greene HL; DAVID Investigators. Percent right ventricular pacing predicts outcomes in the DAVID trial. Heart Rhythm. 2005 Aug;2(8):830-4. doi: 10.1016/j.hrthm.2005.05.015. PMID 16051118
- [Background] Steinberg JS, Fischer A, Wang P, Schuger C, Daubert J, McNitt S, Andrews M, Brown M, Hall WJ, Zareba W, Moss AJ; MADIT II Investigators. The clinical implications of cumulative right ventricular pacing in the multicenter automatic defibrillator trial II. J Cardiovasc Electrophysiol. 2005 Apr;16(4):359-65. doi: 10.1046/j.1540-8167.2005.50038.x. PMID 15828875
- [Background] Vijayaraman P, Bordachar P, Ellenbogen KA. The Continued Search for Physiological Pacing: Where Are We Now? J Am Coll Cardiol. 2017 Jun 27;69(25):3099-3114. doi: 10.1016/j.jacc.2017.05.005. PMID 28641799
- [Background] Boriani G, Pieragnoli P, Botto GL, Puererfellner H, Mont L, Ziacchi M, Manolis AS, Gulizia M, Tukkie R, Landolina M, Ricciardi G, Cicconelli M, Grammatico A, Biffi M. Effect of PR interval and pacing mode on persistent atrial fibrillation incidence in dual chamber pacemaker patients: a sub-study of the international randomized MINERVA trial. Europace. 2019 Apr 1;21(4):636-644. doi: 10.1093/europace/euy286. PMID 30649270
- [Background] Curtis AB, Worley SJ, Chung ES, Li P, Christman SA, St John Sutton M. Improvement in Clinical Outcomes With Biventricular Versus Right Ventricular Pacing: The BLOCK HF Study. J Am Coll Cardiol. 2016 May 10;67(18):2148-2157. doi: 10.1016/j.jacc.2016.02.051. PMID 27151347
- [Background] Beck H, Curtis AB. Right Ventricular Versus Biventricular Pacing for Heart Failure and Atrioventricular Block. Curr Heart Fail Rep. 2016 Oct;13(5):230-236. doi: 10.1007/s11897-016-0299-3. PMID 27553893
- [Background] Sharma PS, Vijayaraman P, Ellenbogen KA. Permanent His bundle pacing: shaping the future of physiological ventricular pacing. Nat Rev Cardiol. 2020 Jan;17(1):22-36. doi: 10.1038/s41569-019-0224-z. Epub 2019 Jun 27. PMID 31249403
- [Background] Vijayaraman P, Chung MK, Dandamudi G, Upadhyay GA, Krishnan K, Crossley G, Bova Campbell K, Lee BK, Refaat MM, Saksena S, Fisher JD, Lakkireddy D; ACC's Electrophysiology Council. His Bundle Pacing. J Am Coll Cardiol. 2018 Aug 21;72(8):927-947. doi: 10.1016/j.jacc.2018.06.017. PMID 30115232
- [Background] Keene D, Arnold AD, Jastrzebski M, Burri H, Zweibel S, Crespo E, Chandrasekaran B, Bassi S, Joghetaei N, Swift M, Moskal P, Francis DP, Foley P, Shun-Shin MJ, Whinnett ZI. His bundle pacing, learning curve, procedure characteristics, safety, and feasibility: Insights from a large international observational study. J Cardiovasc Electrophysiol. 2019 Oct;30(10):1984-1993. doi: 10.1111/jce.14064. Epub 2019 Aug 2. PMID 31310403
- [Background] Jastrzebski M, Moskal P, Bednarek A, Kielbasa G, Czarnecka D. His-bundle pacing as a standard approach in patients with permanent atrial fibrillation and bradycardia. Pacing Clin Electrophysiol. 2018 Nov;41(11):1508-1512. doi: 10.1111/pace.13490. Epub 2018 Sep 19. PMID 30192005
- [Background] Gu M, Hu Y, Hua W, Niu H, Chen X, Cai M, Zhang N, Li H, Zhou X, Zhang S. Visualization of tricuspid valve annulus for implantation of His bundle pacing in patients with symptomatic bradycardia. J Cardiovasc Electrophysiol. 2019 Oct;30(10):2164-2169. doi: 10.1111/jce.14140. Epub 2019 Aug 31. PMID 31456266
- [Background] Vijayaraman P, Dandamudi G. Anatomical approach to permanent His bundle pacing: Optimizing His bundle capture. J Electrocardiol. 2016 Sep-Oct;49(5):649-57. doi: 10.1016/j.jelectrocard.2016.07.003. Epub 2016 Jul 11. PMID 27457727
- [Background] Ponnusamy SS, Arora V, Namboodiri N, Kumar V, Kapoor A, Vijayaraman P. Left bundle branch pacing: A comprehensive review. J Cardiovasc Electrophysiol. 2020 Sep;31(9):2462-2473. doi: 10.1111/jce.14681. Epub 2020 Jul 30. PMID 32681681